CLINICAL TRIAL: NCT06003088
Title: A Randomized, Open-label, Two-Way Crossover Study to Evaluate Relative Bioavailability and Pharmacodynamics of Two Doses of HSK7653 in Healthy Volunteers
Brief Title: Relative Bioavailability and Pharmacodynamics of HSK7653 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HSK7653-105
Record Dates: First submitted 2023-01-11; First posted 2023-08-21 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HSK7653(5mg) Sequence A(Formulation A + Formulation B) (Experimental): Participants will receive a single oral dose of treatment 1: Formulation A followed by a washout period of at least 36 days from first dose of HSK7653(5mg). After the washout period, participants will receive a single oral dose of Treatment 2: HSK7653(5mg) Formulation B.
  Interventions: Drug: HSK7653(5mg)
- HSK7653(5mg) Sequence B(Formulation B + Formulation A) (Experimental): Participants will receive a single oral dose of treatment 1: Formulation B followed by a washout period of at least 36 days from first dose of HSK7653(5mg). After the washout period, participants will receive a single oral dose of Treatment 2: HSK7653(5mg) Formulation A.
  Interventions: Drug: HSK7653(5mg)
- HSK7653(25mg) Sequence A(Formulation A + Formulation B) (Experimental): Participants will receive a single oral dose of treatment 1: Formulation A followed by a washout period of at least 36 days from first dose of HSK7653(25mg). After the washout period, participants will receive a single oral dose of Treatment 2: HSK7653(25mg) Formulation B.
  Interventions: Drug: HSK7653(25mg)
- HSK7653(25mg) Sequence B(Formulation B + Formulation A) (Experimental): Participants will receive a single oral dose of treatment 1: Formulation B followed by a washout period of at least 36 days from first dose of HSK7653(25mg). After the washout period, participants will receive a single oral dose of Treatment 2: HSK7653(25mg) Formulation A.
  Interventions: Drug: HSK7653(25mg)

INTERVENTIONS:
Drug: HSK7653(5mg) — Participants will receive a single oral dose of HSK7653(5mg) Formulation A Or a single oral dose of HSK7653(5mg) Formulation B on Day 1 Period 1. Depending on what Formulation was received on Day 1 Period 1, participants will receive either a single oral dose of HSK7653(5mg) Formulation A Or a single oral dose of HSK7653(5mg) Formulation B on Day 1 of Period 2. Each period lasts for 15 days.
  Other Names: HSK7653
  Arms: HSK7653(5mg) Sequence A(Formulation A + Formulation B); HSK7653(5mg) Sequence B(Formulation B + Formulation A)
Drug: HSK7653(25mg) — Participants will receive a single oral dose of HSK7653(25mg) Formulation A Or a single oral dose of HSK7653(25mg) Formulation B on Day 1 Period 1. Depending on what Formulation was received on Day 1 Period 1, participants will receive either a single oral dose of HSK7653(25mg) Formulation A Or a single oral dose of HSK7653(25mg) Formulation B on Day 1 of Period 2. Each period lasts for 15 days.
  Other Names: HSK7653
  Arms: HSK7653(25mg) Sequence A(Formulation A + Formulation B); HSK7653(25mg) Sequence B(Formulation B + Formulation A)

SUMMARY:
To investigate the relative bioavailability of HSK7653(5mg) given as formulation A versus formulation B.

To investigate the relative bioavailability of HSK7653(25mg) given as formulation A versus formulation B.

To investigate safety and pharmacodynamics of two doses of HSK7653 in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female subjects, age ≥18 years old，with appropriate sex ratio；
2. A total body weight ≥40 kg for females and ≥50 kg for males；BMI of 19 to 26 kg/m^2(inclusive);
3. Subjects(and their partners) volunteered to use effective physical contraception, had no plans to have children or donate sperm/eggs from 14 days before the first dose to 6 months after the last dose;
4. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.

Exclusion Criteria:

1. Subjects who are allergic to two or more medicine, foods or pollens or have a history of allergy to the investigational product and the related compounds;
2. Have a history of severe unconscious hypoglycemia；
3. Clinical evidence or history of any of the following diseases:

   * Inflammatory bowel disease, gastritis, ulcers, bile duct stones, or gastrointestinal bleeding
   * Major gastrointestinal surgery (e.g., gastrectomy, gastrostomy, or enterectomy)
   * Pancreatic injury or pancreatitis
   * Abnormal liver function tests (such as ALT, AST, serum bilirubin) , indicating liver disease or liver injury
   * Renal insufficiency
   * Urinary tract obstruction or difficulty in bladder emptying;
4. Evidence or history of chronic or serious diseases of the blood system, circulatory system, digestive system, urinary system, respiratory system, nervous system, immune system, endocrine system, mental disorders, metabolic disorders, or any other diseases that may affect the results of the study;
5. Serious trauma and surgery within 3 month prior to Screening;
6. Use of vaccines within 1 month prior to dosing;
7. Use of prescription within 1 month prior to dosing，or use of nonprescription drugs（i.e. vitamins and herbal medicines）within 14 days prior to dosing;
8. Participation in another trial with an investigational drug or instrument within 3 months prior to dosing and for the duration of the study;
9. History of regular alcohol consumption exceeding 14 drinks/week (1 drink = 150 mL of wine or 360 mL of beer or 45 mL of hard liquor) within 6 months of Screening.
10. Use of alcohol during the trial,or have a positive result for alcohol breath test;
11. Smoking ≥5 cigarettes per day within 3 months prior to Screening;
12. Blood donation or loss of blood for≥ 400 mL or received blood transfusion or use of blood products within 3 months prior to Screening, or blood donation program for the duration of the study and for 1 month after the trial；
13. Drinking excessive amounts of tea, coffee, and/or caffeinated beverages daily (average more than 8 cups per day,1 cup =250 mL) within 3 months prior to Screening;
14. Use of grapefruit, pomelo, dragon fruit, mango and other fruits or related products that may affect metabolic enzymes within 7 days prior to dosing;
15. Use of products containing alcohol within 48 hours prior to dosing and for the duration of the study;
16. Smoking or using any tobacco product within 48 hours prior to dosing and for the duration of the study;
17. Strenuous activities within 48 hours prior to dosing;
18. Use of chocolate, food or beverages containing caffeine or xanthine within 48 hours prior to dosing;
19. History of drug abuse or drug dependence;
20. Human immunodeficiency virus (HIV) antibody, hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, or Treponema pallidum antibody (TPPA) has a positive result;
21. Any clinically significant physical examination, vital signs, electrocardiogram or clinical laboratory measurement abnormalities during screening, or Screening 12-lead ECG demonstrating QT interval >440 msec for males and >420 msec for females,or FPG< 3.9mmol/L or > 6.1mmol/L;
22. Pregnant or lactating women, or female subjects whose pregnancy test results are positive;
23. Lactose intolerant；
24. Subjects who have a history of fainting needles and blood, or who cannot tolerate venipuncture blood sampling;
25. Difficulty in swallowing tablets and capsules;
26. Special dietary requirements (e.g. vegetarians) or cannot follow a uniform diet during the trial;
27. Unable to cooperate to complete the study due to other reasons, or in the judgment of the investigator, would make the subject inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2022-08-12 (Actual); Study Completion 2022-09-09 (Actual)

PRIMARY OUTCOMES:
Relative bioavailability (F) | Pre-dose，0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168 and 336 hours post-dose.
  To Evaluate Relative Bioavailability (F) of Two Doses of HSK7653 in Healthy Volunteers.
  Relative bioavailability of HSK7653(5mg) given as formulation A versus formulation B=AUC(0-t)(HSK7653(5mg) Formulation A)/AUC(0-t)(HSK7653(5mg) Formulation B).
  Relative bioavailability of HSK7653(25mg) given as formulation A versus formulation B=AUC(0-t)(HSK7653(25mg) Formulation A)/AUC(0-t)(HSK7653(25mg) Formulation B).
AUC(0-t) | Pre-dose，0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168 and 336 hours post-dose.
  The pharmacokinetic parameters of HSK7653 in plasma
AUC(0-∞) | Pre-dose，0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168 and 336 hours post-dose.
  The pharmacokinetic parameters of HSK7653 in plasma
Cmax | Pre-dose，0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168 and 336 hours post-dose.
  The pharmacokinetic parameters of HSK7653 in plasma
Tmax | Pre-dose，0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168 and 336 hours post-dose.
  The pharmacokinetic parameters of HSK7653 in plasma
t1/2 | Pre-dose，0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168 and 336 hours post-dose.
  The pharmacokinetic parameters of HSK7653 in plasma
λz | Pre-dose，0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168 and 336 hours post-dose.
  The pharmacokinetic parameters of HSK7653 in plasma
Vd/F | Pre-dose，0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168 and 336 hours post-dose.
  The pharmacokinetic parameters of HSK7653 in plasma
CL/F | Pre-dose，0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168 and 336 hours post-dose.
  The pharmacokinetic parameters of HSK7653 in plasma

SECONDARY OUTCOMES:
The Safety of HSK7653 | From First dose until Follow up visit, assessed up to 3 months.
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0.
AUEC(0-last) | Pre-dose，0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168 and 336 hours post-dose.
  The pharmacodynamic parameters of HSK7653 in plasma
ECmax | Pre-dose，0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168 and 336 hours post-dose.
  The pharmacodynamic parameters of HSK7653 in plasma
ETmax | Pre-dose，0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168 and 336 hours post-dose.
  The pharmacodynamic parameters of HSK7653 in plasma
DPP-4(WAI-2W) | Pre-dose，0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168 and 336 hours post-dose.
  The pharmacodynamic parameters of HSK7653 in plasma

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Liaoning University of Traditional Chinese Medicine, Shenyang, Liaoning, China